CLINICAL TRIAL: NCT04550208
Title: Biomechanical Analysis of Different Landing Manoevres in Volleyball and Basketball Players
Brief Title: Biomechanical Analysis of Different Landing Manoevres
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000525
Record Dates: First submitted 2020-08-24; First posted 2020-09-16 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2020-08

CONDITIONS: Landing Biomechanics
Keywords: landing; biomechanics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy basketball or volleyball players: Basketball and volleyball players Landing biomechanics of different landing tasks is investigated in a population of volleyball and basketball players
  Interventions: Other: 3D analysis of different landing tasks

INTERVENTIONS:
Other: 3D analysis of different landing tasks — General as well as more sport-specific landing tasks are investigated with 3D analysis by using an opto-electronic system

SUMMARY:
In this study, three-dimensional biomechanics , by means of lower limb joint angles and moments (opto-electronic system with synchronised force plate), of different landing manoevres will be compared in a population of basketball and volleyball players.

DETAILED DESCRIPTION:
In this study, three-dimensional biomechanics , by means of lower limb joint angles and moments (opto-electronic system with synchronised force plate), of different landing manoevres will be compared in a population of basketball and volleyball players. General as well as more sport-specific jumps will be performed in this study.

ELIGIBILITY:
Inclusion Criteria:

* volleyball and basketball players
* male

Exclusion Criteria:

* history or surgery of the lower extremities
* history of fractures of the lower extremities

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volleyball and basketball players
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
External knee joint moments | comparison between 2 different test moments separated by one week
  Knee joint moments will be extracted with an opto-electronic system and synchronised force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Camilla De Bleecker, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided